CLINICAL TRIAL: NCT03097653
Title: New Invited Women to Breast Cancer Screening: a Multi-centre, Longitudinal, Controlled, Randomised Study on a Decision-aid to Support Informed Choice
Brief Title: Decision-aid on Breast Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRFMN-AIRC-6901
Record Dates: First submitted 2017-03-16; First posted 2017-03-31 (Actual); Results first posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Breast Cancer
Keywords: breast cancer screening; mammography; decision-aid; informed choice; National Cancer Screening Program
MeSH Terms: conditions — Breast Neoplasms | interventions — Decision Support Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decision-aid (Experimental)
  Interventions: Other: Decision-aid
- Standard information (Active Comparator)
  Interventions: Other: Standard information

INTERVENTIONS:
Other: Decision-aid — Web platform with a multilevel information and an aid for the decision to be taken. The content is splitted in 16-20 screens; each screen contains the answer to a common question (i.e. What is mammography screening? What are its benefits and harms? What results can be expected from the participation to mammography screening? What is breast cancer?). The information covers also controversial topics as overdiagnosis, overtreatment and the disagreement among scientists about harms and benefits' quantification.
  Arms: Decision-aid
Other: Standard information — Web platform with a standard brochure. This standard brochure represents a combination of the best information available from the three participate centre' brochures.
  Arms: Standard information

SUMMARY:
The present study aim to assess the effect of an interactive web decision aid on informed choice - measured via knowledge, attitudes and intentions concerning breast cancer screening - comparing the decision aid with a standard information provided via web.

DETAILED DESCRIPTION:
Breast cancer is the most common cancer in women. In Italy, women are invited to a population-based mammography screening programme for the first time at the age of 45 or 50 years. Results from randomised controlled trials, observational studies, and systematic reviews continuously fuel the debate on the balance on benefits (reducing breast cancer mortality) and harms (overdiagnosis, overtreatment) of mammography screening. Physicians, policy makers, as well as laypeople or patient associations agree on the need to inform women about the potential benefits and harms in order to allow an aware decision process. Decision aids are an effective way to support lay people in their decisions about health.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 45-69, according to the target age of the screening centres involved;
* New invited women in mammography screening programme.

Exclusion Criteria:

* None

Ages: 45 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1001 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-04-20 (Actual); Study Completion 2019-04-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- Italy (7):
  - Screening Unit, Cancer Prevention and Research Institute - ISPO, Florence
  - UOC Medicina Preventiva delle Comunità - Screening, Milan
  - IRCCS-Istituto di Ricerche Farmacologiche Mario Negri, Milan
  - U.O. Centro Gestionale Screening, Azienda Sanitaria Provinciale di Palermo, Palermo
  - Centro Screeening - AUSL Reggio Emilia, Reggio Emilia
  - CPO Piemonte, Torino
  - SSD Epidemiologia e Screening - CPO Piemonte - AOU Città della Salute e della Scienza, Torino

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Roberto A, Colombo C, Candiani G, Giordano L, Mantellini P, Paci E, Satolli R, Valenza M, Mosconi P. Personalised informed choice on evidence and controversy on mammography screening: study protocol for a randomized controlled trial. BMC Cancer. 2017 Jun 19;17(1):429. doi: 10.1186/s12885-017-3428-9. PMID 28629329
- [Result] Roberto A, Colombo C, Candiani G, Satolli R, Giordano L, Jaramillo L, Castagno R, Mantellini P, Falini P, Carnesciali E, Valenza M, Costa L, Campari C, Caroli S, Faggiano RC, Orione L, Belmessieri B, Marchio V, Deandrea S, Silvestri A, Luciano D, Paci E, Mosconi P. A dynamic web-based decision aid to improve informed choice in organised breast cancer screening. A pragmatic randomised trial in Italy. Br J Cancer. 2020 Sep;123(5):714-721. doi: 10.1038/s41416-020-0935-2. Epub 2020 Jun 17. PMID 32546834

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Date of first enrollment: September 2017 Date of last invitation: 31 December 2018 End of study: April 2019
Period: Overall Study
Arm/Group | Decision-aid | Standard Information
Started | 472 | 529
Completed | 472 | 529
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Decision-aid | Standard Information | Total
Number analyzed (Participants) | 472 | 529 | 1001
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.0 (3.0) | 49.2 (3.3) | 49.1 (3.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 472 | 529 | 1001
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Italian | 458 | 506 | 964
  Other | 12 | 20 | 32
  Missing | 2 | 3 | 5
Marital status [Number; unit: participants]
  Unmarried | 60 | 61 | 121
  Married or cohabitant | 342 | 386 | 728
  Separated or divorced | 62 | 73 | 135
  Widowed | 6 | 6 | 12
  Missing | 2 | 3 | 5
Education [Number; unit: participants]
  Elementary | 2 | 4 | 6
  Lower middle | 69 | 71 | 140
  Higher middle | 234 | 272 | 506
  Degree | 156 | 170 | 326
  Other | 9 | 9 | 18
  Missing | 2 | 3 | 5
Employment status [Number; unit: participants]
  Paid work | 366 | 425 | 791
  No paid work | 104 | 101 | 205
  Missing | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adequate Knowledge
Description: Knowledge will be measured using a questionnaire structured in 13 questions with multiple choice answers, with 2 to 4 options. Ten questions will be qualitative and 3 will be numerical. A score of 8 out of 13 (about 60%) or higher would be considered "adequate knowledge".
Time Frame: 7-10 days
Measure: Number; unit: participants
Arm/Group | Decision-aid | Standard Information
Number analyzed (Participants) | 472 | 529
participants | 236 | 218

2. Primary Outcome: Attitude
Description: Attitude will be measured through a scale of 6 items with 5 response options from 1 to 5, with a total score from 6 to 30. The investigators set the threshold for a positive attitude at 24 and consequently the score <24 point a negative attitude.
Time Frame: 7-10 days
Population: Positive attitude
Measure: Number; unit: participants
Arm/Group | Decision-aid | Standard Information
Number analyzed (Participants) | 472 | 529
participants | 432 | 489

3. Primary Outcome: Intention
Description: Intention will be measured using 1 item with 5 responses: Definitely will, Likely to, Unsure, Not likely to, Definitely will not. The investigators classified "definitely will" and "likely to" as positive intentions.
Time Frame: 7-10 days
Population: Positive intention
Measure: Number; unit: participants
Arm/Group | Decision-aid | Standard Information
Number analyzed (Participants) | 472 | 529
participants | 460 | 500

4. Secondary Outcome: Participation Rate to the Breast Cancer Screening Programme
Description: Participation rate to the breast cancer screening programme will be assessed as a percentage of participants who actually participate, both in intervention and in the control group.
Time Frame: 15-60 days
Population: Participants who had already had a mammogram in the past 6 months were excluded from this dataset.
Measure: Number; unit: percentage of participants
Arm/Group | Decision-aid | Standard Information
Number analyzed (Participants) | 447 | 501
percentage of participants | 84.1 | 83.0

5. Secondary Outcome: Satisfaction With the Information Measured Using 8 Items With Three Points Scale
Description: Satisfaction with the given information will be measured using 8 items with three points scale.
Time Frame: 7-10 days
Population: Satisfaction with the information given (intervention and control group) will be measured using 8 items regarding length, quantity, clarity, balance, helpfulness in making decision and women willingness to recommend it to other women with three points scale
Measure: Number; unit: participants
Arm/Group | Decision-aid | Standard Information
Number analyzed (Participants) | 472 | 529
participants
  Too much | 17 | 6
  Too little | 19 | 31
  Fair | 432 | 480
  Missing | 4 | 12

6. Secondary Outcome: Number of Click on the Homepage
Description: Number of click on the Homepage will be assessed trough Pickwick software.
Time Frame: Through study completion, an average of 10 days
Measure: Number; unit: clicks
Arm/Group | Decision-aid | Standard Information
Number analyzed (Participants) | 472 | 529
clicks | 514 | 334

7. Secondary Outcome: Number of Times Web Platforms Were Accessed
Description: Number of Times Web Platforms were Accessed assessed trough Pickwick software
Time Frame: Through study completion, an average of 10 days
Measure: Mean (Standard Deviation); unit: number of access
Arm/Group | Decision-aid | Standard Information
Number analyzed (Participants) | 472 | 529
number of access | 1.1 (0.3) | 1.0 (0.1)

8. Secondary Outcome: Number of Pages Visited on the Web Platforms
Description: Number of Pages Visited on the Web Platforms on the web decision aid assessed trough Pickwick software.
Time Frame: Through study completion, an average of 10 days
Population: This outcome has been measured only for the interventional arm (Web Decision-aid is splitted in 16-20 screens) because the control arm was just a single webpage.
Measure: Mean (Standard Deviation); unit: Number of pages
Arm/Group | Decision-aid
Number analyzed (Participants) | 472
Number of pages | 4.8 (4.2)

9. Secondary Outcome: Number of Participants With Decisional Conflict Using Decisional Conflict Scale-SURE Version
Description: Decisional conflict will be assessed using the validated and widely used Decisional Conflict Scale-SURE version, consisted in four-item scale.
Time Frame: 7-10 days
Measure: Number; unit: participants
Arm/Group | Decision-aid | Standard Information
Number analyzed (Participants) | 472 | 529
participants
  Decisional conflict (score ≥3) | 68 | 102
  No decisional conflict | 404 | 427

ADVERSE EVENTS:
Time Frame: The aim of this study is the efficacy of a decision-aid on mammography screening. This is not a pharmacological trial, enrolled patients have access to two different kind of web information. Therefore the safety was not considered in this trial and none of the participating women can be considered at risk of adverse effects.
Description: The aim of this study is the efficacy of a decision-aid on mammography screening. This is not a pharmacological trial, enrolled patients have access to two different kind of web information. Therefore the safety was not considered in this trial and none of the participating women can be considered at risk of adverse effects. .
Arm/Group | Decision-aid | Standard Information
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The response rate was lower than expected, and there were about 50% dropouts. We invited more women than expected (21,014 versus 8,160). This high proportion of dropouts could be also due to scarce attention of women to comply with this type of study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-01): https://cdn.clinicaltrials.gov/large-docs/53/NCT03097653/Prot_SAP_000.pdf